

INSTITUTIONAL REVIEW BOARD (IRE) SMAIRH ZAYED PEDERAL POSTGRADUTE MEDICAL INSTITUTE, OF THE DESCRIPTION OF THE STATE



Ret. No. 52+00 flofexton / 0040/2020

Dated: 13 . 64 1616

IRB ID:

IRB APPPROVAL LETTER

Project:

SZMC / IRB / External / Ph.D / 210 / 2020

EFFECTIVENESS OF THINKING HEALTHY PROGRAM FOR PREVENTION OF ANTENATAL DEPRESSION TO IMPROVE MATERNAL HEATH,

Investigator:

Miss. Quratulain (Student Ph.D Public Health)

Department:

Institute of Social & Cultural Studies, University of the Punjah, Lahore

Supervisor:

Dr. Javaria Saleem

Director Institute:

Prof. Dr. Rubeena Zakar

Data Approval:

13.03.2020

Your request for collection of data from the outdoor pregnant women visited to Gynecology & Obstetric Department of Shaikh Zayed Hospital, Lahore is discussed and reviewed by the member of subcommittee, Institutional Review Board (IRB). You are allowed to collect data for your research.

You are directed to follow the rules and regulations as mentioned in your undertaking form,

ROF, DR. MUHAMMAD SUHALL

Beech

Chairman IRB, Institutional Review Board Shaikh Zayed Medical Complex, Lahore

PROF. DR. MUHAMMAD SUHAIL

Chairman, Institutional Review Board Bhaikh Zayed Medical Complex, Lahore

This IRB approval is issued subject to the following conditions:-

- A signed personal declaration of responsibility.
- If the research protocol approved by the IRB changes significantly which alters the nature of 2. the study, a new application for IRB clearance must be submitted.
- It is the principal investigator's responsibility to retain all the necessary forms and informed 3. consent for future reference.

C.C

1. The Deputy Dean, SZPGMI, Lahore

#### **Thinking Healthy Program**

Asalam-u-Alaikum,

#### **Introduction:**

Sheikh Zyed Hospital's Obstetrics and Gynaecology department welcomes you in Program, which aims to support the mental and physical health of pregnant mothers and their baby. We invite you to take part in this program but before participating, it is important for you to know the purpose of this program.

### The purpose of the Program:

In Pakistan, pregnant women frequently face different problems such as stress, anxiety and restlessness. During pregnancy, the presence of stress and anxiety can adversely affect the health of both mother and baby. A special psychosocial based training will be delivered under the supervision of specialists at Sheikh Zyed Hospital's gynaecology department.

#### Why have I been chosen?

This program is for all mothers. You are selected for this program because you will become a mother soon and in our assessment phase we have seen signs of pregnancy related anxiety in you. Therefore, we will ask you some questions regarding your health and your child's health

#### Do I have to take part in this study?

It is entirely your decision whether you want to take part in the study or not. If you decide to take part, but later change your mind you are free to withdraw at any time. Your decision not to take part in the study or withdrawal at any stage will not affect the care you receive now or in the future.

#### How often will I be interviewed?

In addition to the questions about feelings and emotions as well as your family life, you will be interviewed three times by our research team during the duration of the study. This will happen at your first trimester, 3<sup>rd</sup> trimester and 6 weeks after the birth of your baby. The research team can conduct the interview in hospital. The research team consists of female researchers who will ask questions about your emotions, well-being and difficulties you are experiencing concerning your health.

#### What are the possible benefits of taking part?

Purpose of this program is to betterment of mother and child health. By participating in this study, you

will have the opportunity to share your relevant experiences, which may feel beneficial to you and beneficial for other mothers.

### What are the possible disadvantages and risks of taking part?

This study does not involve any physical risks or harm. However sometimes, talking about your experiences and feelings may be difficult and can cause you to be upset. If you feel distressed you will be offered to speak to a counselor. Furthermore, you have the right to refuse to answer a question if you don't feel comfortable answering and can stop the interview at any time if you feel stressed, or simply do not wish to continue.

#### Will my information be kept confidential?

All the information I will collect from you will be strictly confidential. Information will be stored, in a locked cabinet, in our main office, with access available to only research team members. The information will be stored for five years, following the end of the program in 2022, before being destroyed. We might use the information for writing papers or doing presentations at conferences. However, all information will be made anonymous and your identity will not be revealed to anyone at any stage.

Confidentiality will only be breached if there is serious risk of harm to you or to others. Under these conditions we will inform the appropriate health professional so that urgent help can be provided to you.

# Consent (baseline)

## Please initial all boxes

| 1. | I confirm that I have read and understood the information the attached document | Yes | No |
|---|---|---|---|
| | for the study described above. I have had the opportunity to consider the | | |
| | information, ask questions and have had these answered satisfactorily. | | |
| 2. | My participation is voluntary and I am free to withdraw at any time without | Yes | No |
| | giving any reason, without my medical care or legal rights being affected. | | |
| 3. | Information will be kept confidential and I give permission to specialist of this | Yes | No |
| | program to have access to my medical records in case of any need. | | |
| 4. | I agree to take part in the program. | Yes | No |

| Name of participant | Date | Signature | |
|---|---|---|---|
| Ask the participarticipant's parent) is unable to | | pression" in this box if the particip | pant (or |
| Name of person taking consent | Date | Signature | |